CLINICAL TRIAL: NCT02612935
Title: An Observational Pilot Study of Lumosity Computerized Cognitive Training in Subjects With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Lumos Labs, Inc. (Industry)
Collaborators: Dignity Health (Other)
Responsible Party: Sponsor
Other Study IDs: LL009 - MS ACHIEVEMENT STUDY
Record Dates: First submitted 2015-11-19; First posted 2015-11-24 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Multiple Sclerosis (MS)
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Lumosity — Lumosity offers a suite of online games focused on stimulating cognitive domains of attention, memory, cognitive flexibility, problem solving, and speed of processing. The Lumosity program may be well suited for cognitive remediation in individuals with MS.

SUMMARY:
In collaboration with the Mercy MS Achievement Center, Lumos Labs is proposing an open-label, 12-month pilot study of computerized cognitive training as part of the cognitive wellness program in order to evaluate (1) the user experience of Lumosity in individuals with MS, and (2) the efficacy of Lumosity for improving cognitive outcomes in individuals with MS.

DETAILED DESCRIPTION:
Approximately 50 current members of the Mercy MS Achievement Center will be provided with 12-month premium access Lumosity accounts. Study participants must be ≥18 years of age, and currently members of the Achievement Center participating in the cognitive wellness program. Those who consent will be provided with an account activation code and instructed on how to sign up for Lumosity.

Upon creating an account, users would be asked to complete a short demographic survey (Information About You, which includes age, sex, race/ethnicity, education, occupation) and two additional short surveys: a Computer Experience Questionnaire and a Perceptions of Brain Training questionnaire. In addition, participants will be assessed with the Montreal Cognitive Assessment (MOCA), and be directed to take the Brain Performance Test (on a laptop or desktop computer) within the first 7 days of creating their account. If not conducted within the previous 3 months, participants would also be required to have the following assessments at baseline (i.e., within the first 7 days): Multiple Sclerosis Neuropsychological Questionnaire (MSNQ), Multiple Sclerosis Impact Scale-29 (MSIS-29), and Beck Depression Inventory (BDI). After one week of using Lumosity, and then every other month for 12 months, participants would be asked to complete a short questionnaire about their experience with Lumosity. Every 3 months, participants would repeat the BPT, MSNQ, and BDI; and every 6 months, they would repeat the MSIS. Finally, at the end of the study, the end of the study they would also repeat the MOCA.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet the following criteria:

1. Signed informed consent
2. 18 years of age or older,
3. English-speaking,
4. Current participants in the MS Achievement Center Cognitive Wellness Program
5. Sufficient physical capacity to use a computer keyboard and mouse
6. Willing and able to use Lumosity at least 3 times per week

Exclusion Criteria:

Participants who meet any of the following criteria will be excluded from participation:

1. Under 18 years of age
2. Are taking medication that may impede cognitive functioning
3. Have other conditions or problems that may preclude regular computer usage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 50 current members of the Mercy MS Achievement Center will be provided with 12-month premium access Lumosity accounts. Study participants must be ≥18 years of age, and currently members of the Achievement Center participating in the cognitive wellness program.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2015-03; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Performance Characteristics and Usability measures of Lumosity, as measured by Self-Report Descriptive Questionnaires | 1 year
  The primary objective is to determine performance characteristics and usability of Lumosity in individuals with MS as measured through qualitative questionnaires.

SECONDARY OUTCOMES:
Efficacy of Lumosity in individuals with MS, as measured with the BPT | Change from baseline as measured at 3, 6, 9 and 12 months
  To determine the efficacy of Lumosity in this study population as measured by change from baseline on the BPT Grand Index score and scaled subtest scores at 3, 6, 9, and 12 months
Efficacy of Lumosity in individuals with MS, as measured with the MSNQ | 1 Year
  To determine the efficacy of Lumosity in this study population as measured by
  • Change from baseline on the MSNQ at 12 months
Efficacy of Lumosity in individuals with MS, as measured with the MOCA | 1 Year
  To determine the efficacy of Lumosity in this study population as measured by
  • Change from baseline on the MOCA at 12 months
Efficacy of Lumosity in individuals with MS, as measured with the MSIS-29. | 1 Year
  To determine the efficacy of Lumosity in this study population as measured by
  • Change from baseline on the MSIS-29 at 12 months
Efficacy of Lumosity in individuals with MS, as measured with the BDI. | 1 Year
  To determine the efficacy of Lumosity in this study population as measured by
  • Change from baseline on the BDI at 12 months
Engagement - as measured by number of unique days played and number of games played | 1 year
  To determine the level of engagement with Lumosity in individuals with MS as measured by number of unique days and number of games played

CONTACTS AND LOCATIONS:
Overall Officials: Brian Hutchinson, Principal Investigator — MS Achievement Center